CLINICAL TRIAL: NCT05485103
Title: A Prospective Study of the Effect of Modified Colonoscopy Bowel Preparation Program on Intestinal Cleaning, Examination and Disease in Patients With Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZS-3300
Record Dates: First submitted 2022-07-05; First posted 2022-08-03 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-06

CONDITIONS: Inflammatory Bowel Diseases
Keywords: modified bowel preparation method; inflammatory bowel disease; risk factors; quality of bowel preparation
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Polyethylene Glycols

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified bowel preparation method group (Experimental): One day before the colonoscopy, only asol (or other intestinal nutrient solution) was taken. On the examination day (4 hours before), 1 bag of polyethylene glycol solution + (2 hours before) glycerin enema 110ml was taken
  Interventions: Drug: Polyethylene Glycols
- Traditional bowel preparation method group (Active Comparator): Low residue diet 2 days before the colonoscopy, take 2 bags of polyethylene glycol solution the night before the examination and 1 bag of which on the examination day (4 hours before)
  Interventions: Drug: Polyethylene Glycols

INTERVENTIONS:
Drug: Polyethylene Glycols — Take asol as total enteral nutrition, and take polyethylene glycols and glycerin enema as bowel preparations
  Other Names: glycerin enema; asol

SUMMARY:
The purpose of this study is to investigate the effect of modified colonoscopy bowel preparation method compared with traditional method on bowel cleansing effect, colonoscopy examination effect and clinical condition of inflammatory bowel disease patients. Risk factors affecting the quality of bowel preparation will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: inflammatory bowel disease (IBD) patients, including ulcerative colitis (UC) and Crohn's disease (CD), have colonic involvement.
* Patients and/or family members can understand the study protocol and are willing to participate in the study and provide informed consent in writing.

Exclusion Criteria:

* The diagnosis is not definite.
* Toxic megacolon, gastrointestinal perforation or other acute abdominal diseases; Patients with gastrointestinal bleeding with unstable vital signs.
* Patients after colon surgery.
* Serious underlying diseases, organ failure, or inability to cooperate with colonoscopy for other reasons.
* Patients can not cooperate with the use of polyethylene glycol or glycerin enema.
* Patients or family members cannot understand the conditions and objectives of this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The quality of bowel preparation evaluated by endoscopists during colonoscopy. | During colonoscopy examination
  The quality of bowel preparation will be evaluated with the Boston bowel preparation scale (BBPS), including the total Boston score (range 0-9, score 8-9 means excellent, 7 means good, less than 7 means bad) and score of per bowel segment (maximum 3).
Number of Participants with increased Disease activity after colonoscopy. | Within 7 days after colonoscopy
  Disease activity will be assessed using C-reactive protein (CRP) measurement, the modified Mayo score in ulcerative colitis and the Crohn's Disease Activity Index score in Crohn's Disease. If the result after colonoscopy was higher than before, the participant may be considered with increased disease activity.

SECONDARY OUTCOMES:
Tolerance score of participants after bowel preparation. | After bowel preparation and before colonoscopy
  Tolerance score is defined range 0-10 (0 means totally intolerant, 10 means feel really good).
Number of Participants who has a record of outpatient or emergency treatment due to aggravation of disease after colonoscopy. | Within 30 days after colonoscopy
  Number of Participants who has a record of outpatient or emergency treatment due to aggravation of disease within 30 days after colonoscopy.
Number of Participants hospitalized because of aggravation of disease after colonoscopy. | Within 30 days after colonoscopy
  Number of Participants who is hospitalized because of aggravation of disease within 30 days after colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Xu, MD, Study Chair — Peking Union Medical College Hospital
Locations (9):
- China (9):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Sixth Hospital, Beijing, Beijing Municipality
  - Heilongjiang Provincial Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The first Hospital of China Medical University, Shenyang, Liaoning
  - The second Affiliated Hospital of Baotou Medical Colledge, Baotou, Neimenggu
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Beijing Rectum Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sultan K, Trindade AJ. Concise Commentary: Is Splitting the Difference? Identifying Risk Factors Associated with Suboptimal Bowel Preparation for Colonoscopy Among IBD Patients. Dig Dis Sci. 2022 Oct;67(10):4602-4603. doi: 10.1007/s10620-022-07533-5. Epub 2022 May 17. No abstract available. PMID 35579796
- [Background] Kim KO, Kim EY, Lee YJ, Lee HS, Kim ES, Chung YJ, Jang BI, Kim SK, Yang CH. Efficacy, safety and tolerability of oral sulphate tablet for bowel preparation in patients with inflammatory bowel disease: A multicentre randomized controlled study. J Crohns Colitis. 2022 Nov 23;16(11):1706-1713. doi: 10.1093/ecco-jcc/jjac080. PMID 35689818
- [Background] Wijnands AM, Te Groen M, Peters Y, Kaptein AA, Oldenburg B, Hoentjen F, Lutgens MWMD. Patients Prioritize a Low-volume Bowel Preparation in Colitis-associated Colorectal Cancer Surveillance: A Discrete Choice Experiment. Inflamm Bowel Dis. 2022 Jul 1;28(7):1053-1060. doi: 10.1093/ibd/izab221. PMID 34487155
- [Background] Reddy P, Mencin A, Lebwohl B. Risk Factors for Suboptimal Bowel Preparation for Colonoscopy in Pediatric Patients. J Pediatr Gastroenterol Nutr. 2021 Jul 1;73(1):e1-e6. doi: 10.1097/MPG.0000000000003114. PMID 33661246
- [Background] Neri B, Scarozza P, Giannarelli D, Sena G, Mossa M, Lolli E, Calabrese E, Biancone L, Grasso E, Di Iorio L, Troncone E, Monteleone G, Paoluzi OA, Del Vecchio Blanco G. Efficacy and tolerability of very low-volume bowel preparation in patients with inflammatory bowel diseases. Eur J Gastroenterol Hepatol. 2021 Jul 1;33(7):977-982. doi: 10.1097/MEG.0000000000002167. PMID 34034275
- [Background] Maida M, Morreale GC, Sferrazza S, Sinagra E, Scalisi G, Vitello A, Vettori G, Rossi F, Catarella D, Di Bartolo CE, Schillaci D, Raimondo D, Camilleri S, Orlando A, Macaluso FS. Effectiveness and safety of 1L PEG-ASC preparation for colonoscopy in patients with inflammatory bowel diseases. Dig Liver Dis. 2021 Sep;53(9):1171-1177. doi: 10.1016/j.dld.2021.04.006. Epub 2021 May 12. PMID 33994129
- [Background] Negreanu L, Voiosu T, State M, Mateescu RB. Quality of colonoscopy preparation in patients with inflammatory bowel disease: retrospective analysis of 348 colonoscopies. J Int Med Res. 2020 Apr;48(4):300060520903654. doi: 10.1177/0300060520903654. PMID 32237946
- [Background] Megna B, Weiss J, Ley D, Saha S, Pfau P, Grimes I, Li Z, Caldera F. Clear liquid diet before bowel preparation predicts successful chromoendoscopy in patients with inflammatory bowel disease. Gastrointest Endosc. 2019 Feb;89(2):373-379.e2. doi: 10.1016/j.gie.2018.09.039. Epub 2018 Oct 16. PMID 30339950
- [Background] Briot C, Faure P, Parmentier AL, Nachury M, Trang C, Viennot S, Altwegg R, Bulois P, Thomassin L, Serrero M, Ah-Soune P, Gilletta C, Plastaras L, Simon M, Dray X, Caillo L, Del Tedesco E, Abitbol V, Zallot C, Degand T, Rossi V, Bonnaud G, Colin D, Morel B, Winkfield B, Danset JB, Filippi J, Amiot A, Attar A, Levy J, Peyrin-Biroulet L, Vuitton L; CLEAN Study Group. Efficacy, Tolerability, and Safety of Low-Volume Bowel Preparations for Patients with Inflammatory Bowel Diseases: The French Multicentre CLEAN Study. J Crohns Colitis. 2019 Sep 19;13(9):1121-1130. doi: 10.1093/ecco-jcc/jjz040. PMID 30785181
- [Background] Spiceland CM, Lodhia N. Endoscopy in inflammatory bowel disease: Role in diagnosis, management, and treatment. World J Gastroenterol. 2018 Sep 21;24(35):4014-4020. doi: 10.3748/wjg.v24.i35.4014. PMID 30254405
- [Background] Martel M, Menard C, Restellini S, Kherad O, Almadi M, Bouchard M, Barkun AN. Which Patient-Related Factors Determine Optimal Bowel Preparation? Curr Treat Options Gastroenterol. 2018 Dec;16(4):406-416. doi: 10.1007/s11938-018-0208-9. PMID 30390208
- [Background] Bezzio C, Andreozzi P, Casini V, Manes G, Saibeni S. Endoscopy for patients affected by inflammatory bowel disease: bowel preparation and sedation. Expert Rev Gastroenterol Hepatol. 2018 Feb;12(2):119-124. doi: 10.1080/17474124.2017.1390430. Epub 2017 Oct 17. PMID 29019424
- [Background] Shobar RM, Velineni S, Keshavarzian A, Swanson G, DeMeo MT, Melson JE, Losurdo J, Engen PA, Sun Y, Koenig L, Mutlu EA. The Effects of Bowel Preparation on Microbiota-Related Metrics Differ in Health and in Inflammatory Bowel Disease and for the Mucosal and Luminal Microbiota Compartments. Clin Transl Gastroenterol. 2016 Feb 11;7(2):e143. doi: 10.1038/ctg.2015.54. PMID 26866392
- [Background] Nett A, Velayos F, McQuaid K. Quality bowel preparation for surveillance colonoscopy in patients with inflammatory bowel disease is a must. Gastrointest Endosc Clin N Am. 2014 Jul;24(3):379-92. doi: 10.1016/j.giec.2014.03.004. Epub 2014 May 6. PMID 24975529
- [Background] Bessissow T, Van Keerberghen CA, Van Oudenhove L, Ferrante M, Vermeire S, Rutgeerts P, Van Assche G. Anxiety is associated with impaired tolerance of colonoscopy preparation in inflammatory bowel disease and controls. J Crohns Colitis. 2013 Dec;7(11):e580-7. doi: 10.1016/j.crohns.2013.04.011. Epub 2013 May 9. PMID 23664621